CLINICAL TRIAL: NCT00219557
Title: A RANDOMIZED PHASE 2 STUDY OF THE ANTI-ANGIOGENESIS AGENT AG-013736 IN COMBINATION WITH GEMCITABINE IN PATIENTS WITH CHEMOTHERAPY-NAIVE ADVANCED PANCREATIC CANCER PRECEDED BY A PHASE 1 PORTION
Brief Title: AG-013736 In Combination With Gemcitabine Versus Gemcitabine Alone For Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061016; 2005-000053-30 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Randomized Phase 2 Study of AG-013736 in Combination with Gemcitabine versus Gemcitabine Alone in Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (Active Comparator)
  Interventions: Drug: Gemcitabine
- Axitinib [AG-013736] plus gemcitabine (Experimental)
  Interventions: Drug: AG-013736; Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 30 minutes IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks
  Arms: Gemcitabine
Drug: AG-013736 — Axitinib (AG-013736) 5 mg tablet orally BID starting from Day 1 of Cycle 1, in cycles of 4 weeks.
  Arms: Axitinib [AG-013736] plus gemcitabine
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 30 minutes IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
  Arms: Axitinib [AG-013736] plus gemcitabine

SUMMARY:
This is a Phase 2 study being conducted at multiple centers in the United States, Europe and Canada. Patients having pancreatic cancer that is locally advanced or that has spread to other parts of the body (i.e., metastatic) are eligible to participate. Patients must have not had any prior systemic treatment for advanced disease. The purpose of the study is to test whether the angiogenesis inhibitor Axitinib [AG-013736] in combination with gemcitabine is an effective treatment for advanced pancreatic cancer vs. gemcitabine alone by overall survival.

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced (localized but surgically unresectable or metastatic) histologically/cytologically proven epithelial cancer of the exocrine pancreas
* no prior therapy for metastatic disease

Exclusion Criteria:

* patients with locally advanced disease who are candidates for radiation therapy.
* uncontrolled brain metastases (a controlled brain metastasis must be previously treated, asymptomatic, and without growth for 4 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-07-05 (Actual); Primary Completion 2008-03-14 (Actual); Study Completion 2008-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (17):
  - East Bay Medical Oncology/Hematology Medical Associates Inc., Antioch, California
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Bay Area Cancer Research Group, Concord, California
  - East Bay Medical Oncology/Hematology Medical Associates, Inc., Concord, California
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Jackson Memorial Hospital & Clinics, Miami, Florida
  - University of Miami Hospital & clinics, Miami, Florida
  - H Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Maine Center for Cancer Medicine and Blood Disorders, Biddeford, Maine
  - Maine Center for Cancer Medicine and Blood Disorders, Brunswick, Maine
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Arch Medical Services, Inc. d/b/a The Center for Cancer Care and Research, St Louis, Missouri
  - Arch Medical Services, Inc. d/b/a The Center for Cancer Care and Research, Washington, Missouri
  - Southeast Nebraska Cancer Center, Southeast Nebraska Hematology and Oncology Consultants, P.C., Lincoln, Nebraska
  - Piedmont Hematology Oncology Association, Winston-Salem, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Universitair Ziekenhuis Gent/Dienst Gastroenterologie, Ghent, Belgium
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM, Hopital Saint-Luc, Montreal, Quebec
- France (4):
  - Service Oncologie Medicale, Saint-Herblain, Saint Herblain Cedex
  - Hopital La Timone, Marseille
  - Hopital de la Pitie Salpetriere, Paris
  - Institut Claudius Regaud, Toulouse
- Medizinische Klinik mit Schwerpunkt Haematologie und Onkologie, Charité-Universitaetsmedizin Berlin, Berlin, Germany
- Italy (2):
  - Fondazione IRCCS, Istituto Nazionale Tumori, Oncologia Medica B, Milan
  - Unita Operativa, Oncologia Medica, Istituto di Medicina Interna e Geriatria, Roma
- Spain (3):
  - Hospital Universitario Vall D´Hebron, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (4):
  - Cancer Research Uk Clinical Centre, Southampton, Hampshire
  - Department of Cancer Studies & Molecular Medicine, Leicester, Leicestershire
  - Western General Hospitals Nhs Trust, Edinburgh
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Spano JP, Chodkiewicz C, Maurel J, Wong R, Wasan H, Barone C, Letourneau R, Bajetta E, Pithavala Y, Bycott P, Trask P, Liau K, Ricart AD, Kim S, Rixe O. Efficacy of gemcitabine plus axitinib compared with gemcitabine alone in patients with advanced pancreatic cancer: an open-label randomised phase II study. Lancet. 2008 Jun 21;371(9630):2101-8. doi: 10.1016/S0140-6736(08)60661-3. Epub 2008 May 29. PMID 18514303
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061016&StudyName=AG-013736%20In%20Combination%20With%20Gemcitabine%20Versus%20Gemcitabine%20Alone%20For%20Patients%20With%20Metastatic%20Pancreatic%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Gemcitabine (Phase 1 Lead-In): Axitinib (AG-013736) 5 milligram (mg) tablet orally twice daily (BID) starting from Day 3 of Cycle 1, in cycles of 4 weeks. Gemcitabine 1000 milligram/square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
- Axitinib + Gemcitabine: Axitinib (AG-013736) 5 mg tablet orally BID starting from Day 1 of Cycle 1, in cycles of 4 weeks. Gemcitabine 1000 mg/m^2 30 minutes IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
Period: Phase 1
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In) | Axitinib + Gemcitabine | Gemcitabine
Started | 8 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Started chemotherapy at other institute | 1 | 0 | 0
Period: Phase 2
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In) | Axitinib + Gemcitabine | Gemcitabine
Started | 0 | 69 | 34
Treated | 0 | 68 | 31
Completed | 0 | 0 | 1
Not Completed | 0 | 69 | 33
Not completed — Lack of Efficacy | 0 | 21 | 15
Not completed — Adverse Event | 0 | 22 | 2
Not completed — Death | 0 | 8 | 2
Not completed — Other | 0 | 8 | 6
Not completed — Withdrawal by Subject | 0 | 9 | 5
Not completed — Treatment not received | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In) | Axitinib + Gemcitabine | Gemcitabine | Total
Number analyzed (Participants) | 8 | 69 | 34 | 111
Age, Customized [Count of Participants; unit: Participants]
  18 years to 44 years | 0 | 2 | 4 | 6
  45 years to 64 years | 5 | 31 | 20 | 56
  Greater than or equal to 65 years | 3 | 36 | 10 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 34 | 18 | 53
  Male | 7 | 35 | 16 | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time in days from randomization to date of death due to any cause. OS was calculated as the death date minus the date of randomization plus 1. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline of Phase 2 to death or until at least 1 year after the randomization of the last participant
Population: Phase 2 intent to treat (ITT) population included all participants randomized with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or a drug different from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 69 | 34
Days | 210 [162 to 308] | 171 [125 to 267]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Gemcitabine; Differences in OS between treatment arms was analyzed by the stratified log-rank test where the stratification factors are Eastern Cooperative Oncology Group (ECOG) performance status (less than or equal to 1 or 2) and extent of disease (locally advanced or metastatic); Test type: Superiority or Other; p = 0.1026, Log Rank — One-sided log-rank test at alpha = 0.1 significance level was used; Hazard Ratio (HR) = 0.758, 95% CI 2-sided [0.490 to 1.170]

2. Secondary Outcome: Dose Confirmation of Axitinib (AG-013736) on Basis of Number of Participants With Dose Limiting Toxicity (DLT)
Description: Dose of axitinib (AG-013736) was confirmed if not more than 1 out of 6 participants experienced a DLT during first cycle. DLT included grade (Gr) 4 neutropenia or thrombocytopenia, greater than or equal to (>=) Gr 3 anemia or non hematological toxicities for >= 7 days (except alopecia) or >= Gr 1 hemoptysis or >=2 gram /24 hours proteinuria or inability to resume background chemotherapy or axitinib (AG-013736) dosing within 14 days of stopping due to treatment related toxicity.
Time Frame: Phase 1 baseline up to Week 4
Population: Phase 1 safety population included all participants who received at least 1 dose of study drug with treatment assignments designated according to actual study treatment received. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: Dose Confirmation of Gemcitabine on Basis of Number of Participants With Dose Limiting Toxicity (DLT)
Description: Dose of gemcitabine was confirmed if not more than 1 out of 6 participants experienced a DLT during first cycle. DLT included grade (Gr) 4 neutropenia or thrombocytopenia, greater than or equal to (>=) Gr 3 anemia or non hematological toxicities for >= 7 days (except alopecia) or >= Gr 1 hemoptysis or >=2 gram /24 hours proteinuria or inability to resume background chemotherapy or axitinib (AG-013736) dosing within 14 days of stopping due to treatment related toxicity.
Time Frame: Phase 1 Baseline up to Week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
participants | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Axitinib (AG-013736)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3.5, 4.5, 9.5, and 12.5 hours (hr) post-dose on Day 15 of Phase 1 Cycle 1
Population: Phase 1 Pharmacokinetic (PK) evaluable population included all ITT participants who completed PK blood sampling on at least 1 day.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
nanogram/milliliter (ng/mL) | 45.08 (34.32)

5. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC (0-24)] of Axitinib (AG-013736)
Description: AUC (0-24) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to 24 hours (0-24).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3.5, 4.5, 9.5, and 12.5 hr post-dose on Day 15 of Phase 1 Cycle 1
Population: Phase 1 PK evaluable population included all participants who completed PK blood sampling on at least 1 day.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
ng*hr/mL | 282.34 (135.27)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Axitinib (AG-013736)
Description: Tmax was based on the actual time points when the samples were collected.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3.5, 4.5, 9.5, and 12.5 hr post-dose on Day 15 of Phase 1 Cycle 1
Population: Phase 1 PK evaluable population included all participants who completed PK blood sampling on at least 1 day.
Measure: Median (Full Range); unit: hr
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
hr | 1.52 [0.50 to 2.20]

7. Secondary Outcome: Plasma Decay Half-life (t1/2) of Axitinib (AG-013736)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3.5, 4.5, 9.5, and 12.5 hr post-dose on Day 15 of Phase 1 Cycle 1
Population: Phase 1 PK evaluable population included all participants who completed PK blood sampling on at least 1 day.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 6
hr | 2.97 (1.95)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Gemcitabine
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 9 and 12 hr after start of infusion on Day 15 of Phase 1 Cycle 1
Population: Phase 1 PK evaluable population included all participants who completed PK blood sampling on at least 1 day. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 5
ng/mL | 27280.0 (12599.1)

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Gemcitabine
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 9 and 12 hr after start of infusion on Day 15 of Phase 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 5
ng*hr/mL | 13656.00 (4142.16)

10. Secondary Outcome: Plasma Decay Half-life (t1/2) of Gemcitabine
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 9 and 12 hr after start of infusion on Day 15 of Phase 1 Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In)
Number analyzed (Participants) | 5
hr | 0.310 (0.028)

11. Secondary Outcome: Population Pharmacokinetics of Axitinib (AG-013736) in Phase 2
Description: Data for this outcome measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Phase 2 Day 1 (Pre-dose), Day 29, Day 57 and then every 8 weeks until disease progression or discontinuation from study or up to 80 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Percentage of Participants With Overall Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non-target). PR are those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum of longest dimensions.
Time Frame: Phase 2 baseline to disease progression or discontinuation from study, assessed every 8 weeks up to 80 weeks
Population: Phase 2 ITT population included all participants randomized with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or a drug different from that to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 69 | 34
Percentage of Participants | 7.2 [2.4 to 16.1] | 2.9 [0.1 to 15.3]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Gemcitabine; Difference in percent of participants with overall response expressed as response rate, was used for calculation of 95% confidence interval (CI); Test type: Superiority or Other; p = 0.661, Fisher Exact; Difference in response rate = 4.3, 95% CI 2-sided [-4.0 to 12.7]

13. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Phase 2 baseline to disease progression or discontinuation from study due to any cause, assessed every 8 weeks up to 80 weeks
Population: Subgroup of participants from Phase 2 ITT population, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 5 | 1
Days | 379 [136 to 379] | 155 [NA to NA] — 95% CI was not estimable because only one participant was evaluable.

14. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in days from randomization to first documentation of objective tumor progression or death due to any cause. PFS was calculated as first event date minus the date of randomization plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Phase 2 baseline until the date of first documented progression or death due to any cause, assessed every 8 weeks up to 80 weeks
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 69 | 34
Days | 116 [109 to 160] | 113 [68 to 205]
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Gemcitabine; Differences in PFS between treatment arms was analyzed by the stratified log-rank test where the stratification factors are ECOG performance status (less than equal to 1 or 2) and extent of disease (locally advanced or metastatic); Test type: Superiority or Other; p = 0.4466, Log Rank — One-sided log-rank test at alpha = 0.1 significance level was used; Hazard Ratio (HR) = 0.9648, 95% CI 2-sided [0.5400 to 1.7300]

15. Secondary Outcome: One Year Survival Probability
Description: One year survival probability was defined as the probability of survival at one year after the date of randomization based on the Kaplan Meier estimate.
Time Frame: Phase 2 baseline to disease progression or death due to any cause or at least 1 year after the first dose for the last participant
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percent chance of survival
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 69 | 34
Percent chance of survival | 36.81 [25.71 to 47.93] | 23.53 [11.48 to 38.01]

16. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score at Day 1 of Every Cycle and End of Study
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning or greater degree of symptoms. Change from baseline=Cycle/Day score minus baseline score.
Time Frame: Phase 2 baseline [Day (D)1 of Cycle (C)1], Day 1 of all subsequent cycles up to Cycle 14 and end of study (EoS).
Population: Phase 2 ITT population was the primary analysis population. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. ''n'' signifies the number of participants evaluable for the respective scale at the respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Axitinib + Gemcitabine: Axitinib (AG-013736) 5 mg tablet orally BID starting from Day 3 of Cycle 1, in cycles of 4 weeks. Gemcitabine 1000 mg/m^2 30 minutes IV infusion on Day 1, 8 and 15 of each cycle, in cycles of 4 weeks.
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 65 | 27
units on a scale
  Global QoL: Baseline | 55.60 (27.18) | 54.32 (21.10)
  Physical Functioning: Baseline | 76.90 (24.73) | 82.22 (14.44)
  Role Functioning: Baseline: number analyzed (Participants) | 65 | 26
  Role Functioning: Baseline | 62.56 (33.21) | 60.26 (35.30)
  Emotional Functioning: Baseline | 67.22 (26.17) | 66.98 (23.96)
  Cognitive Functioning: Baseline | 82.82 (23.93) | 82.10 (19.57)
  Social Functioning: Baseline: number analyzed (Participants) | 65 | 26
  Social Functioning: Baseline | 67.44 (33.00) | 70.51 (29.56)
  Fatigue: Baseline | 43.50 (29.78) | 42.80 (25.73)
  Nausea and Vomiting: Baseline | 19.74 (28.24) | 13.58 (20.17)
  Pain: Baseline | 40.00 (33.31) | 37.04 (31.80)
  Dyspnea: Baseline: number analyzed (Participants) | 64 | 27
  Dyspnea: Baseline | 12.50 (21.82) | 16.05 (26.75)
  Insomnia: Baseline | 31.28 (31.66) | 39.51 (39.26)
  Appetite loss: Baseline | 41.03 (40.30) | 33.33 (34.59)
  Constipation: Baseline | 34.87 (37.93) | 38.27 (38.90)
  Diarrhea: Baseline | 20.00 (27.51) | 16.05 (28.30)
  Financial Difficulties: Baseline: number analyzed (Participants) | 64 | 27
  Financial Difficulties: Baseline | 10.42 (19.59) | 28.40 (41.04)
  Global QoL: Change at C2 D1: number analyzed (Participants) | 49 | 20
  Global QoL: Change at C2 D1 | -5.10 (21.17) | 3.33 (16.97)
  Physical Functioning: Change at C2 D1: number analyzed (Participants) | 51 | 21
  Physical Functioning: Change at C2 D1 | -5.07 (18.85) | 0.95 (16.23)
  Role Functioning: Change at C2 D1: number analyzed (Participants) | 51 | 19
  Role Functioning: Change at C2 D1 | 0.33 (25.93) | 9.65 (29.56)
  Emotional Functioning: Change at C2 D1: number analyzed (Participants) | 52 | 21
  Emotional Functioning: Change at C2 D1 | 3.21 (21.34) | 7.94 (17.77)
  Cognitive Functioning: Change at C2 D1: number analyzed (Participants) | 52 | 21
  Cognitive Functioning: Change at C2 D1 | -3.53 (21.48) | 1.59 (18.93)
  Social Functioning: Change at C2 D1: number analyzed (Participants) | 52 | 20
  Social Functioning: Change at C2 D1 | -4.17 (29.50) | -0.83 (28.85)
  Fatigue: Change at C2 D1: number analyzed (Participants) | 51 | 21
  Fatigue: Change at C2 D1 | 1.42 (21.74) | -8.99 (26.67)
  Nausea and Vomiting: Change at C2 D1: number analyzed (Participants) | 51 | 21
  Nausea and Vomiting: Change at C2 D1 | -5.88 (26.84) | -1.59 (12.81)
  Pain: Change at C2 D1: number analyzed (Participants) | 52 | 21
  Pain: Change at C2 D1 | -9.29 (27.89) | -16.67 (31.62)
  Dyspnea: Change at C2 D1: number analyzed (Participants) | 50 | 21
  Dyspnea: Change at C2 D1 | 9.33 (26.97) | -3.17 (25.61)
  Insomnia: Change at C2 D1: number analyzed (Participants) | 51 | 21
  Insomnia: Change at C2 D1 | -9.15 (28.35) | -19.05 (34.27)
  Appetite loss: Change at C2 D1: number analyzed (Participants) | 51 | 21
  Appetite loss: Change at C2 D1 | -0.65 (35.58) | -14.29 (35.86)
  Constipation: Change at C2 D1: number analyzed (Participants) | 52 | 21
  Constipation: Change at C2 D1 | -9.62 (32.56) | -14.29 (29.00)
  Diarrhea: Change at C2 D1: number analyzed (Participants) | 52 | 21
  Diarrhea: Change at C2 D1 | -1.28 (29.49) | 0.00 (18.26)
  Financial Difficulties: Change at C2 D1: number analyzed (Participants) | 50 | 21
  Financial Difficulties: Change at C2 D1 | 0.67 (19.62) | -4.76 (19.11)
  Global QoL: Change at C3 D1: number analyzed (Participants) | 40 | 15
  Global QoL: Change at C3 D1 | -9.17 (30.36) | 6.67 (15.17)
  Physical Functioning: Change at C3 D1: number analyzed (Participants) | 42 | 15
  Physical Functioning: Change at C3 D1 | -8.13 (21.46) | 3.44 (18.73)
  Role Functioning: Change at C3 D1: number analyzed (Participants) | 42 | 14
  Role Functioning: Change at C3 D1 | -5.56 (27.71) | 13.10 (25.47)
  Emotional Functioning: Change at C3 D1: number analyzed (Participants) | 41 | 15
  Emotional Functioning: Change at C3 D1 | -1.69 (26.80) | 12.22 (19.89)
  Cognitive Functioning: Change at C3 D1: number analyzed (Participants) | 41 | 15
  Cognitive Functioning: Change at C3 D1 | -4.88 (24.79) | 2.22 (16.51)
  Social Functioning: Change at C3 D1: number analyzed (Participants) | 41 | 15
  Social Functioning: Change at C3 D1 | -4.07 (32.66) | 5.56 (24.93)
  Fatigue: Change at C3 D1: number analyzed (Participants) | 42 | 14
  Fatigue: Change at C3 D1 | 7.41 (28.61) | -8.73 (26.57)
  Nausea and Vomiting: Change at C3 D1: number analyzed (Participants) | 42 | 13
  Nausea and Vomiting: Change at C3 D1 | -4.37 (29.00) | -2.56 (16.45)
  Pain: Change at C3 D1: number analyzed (Participants) | 42 | 15
  Pain: Change at C3 D1 | -6.75 (33.75) | -23.33 (30.08)
  Dyspnea: Change at C3 D1: number analyzed (Participants) | 41 | 14
  Dyspnea: Change at C3 D1 | 3.25 (27.69) | -7.14 (19.30)
  Insomnia: Change at C3 D1: number analyzed (Participants) | 42 | 14
  Insomnia: Change at C3 D1 | -10.32 (34.13) | -11.90 (38.36)
  Appetite loss: Change at C3 D1: number analyzed (Participants) | 42 | 13
  Appetite loss: Change at C3 D1 | 11.11 (39.42) | -5.13 (29.96)
  Constipation: Change at C3 D1: number analyzed (Participants) | 41 | 15
  Constipation: Change at C3 D1 | -10.57 (32.86) | -13.33 (35.19)
  Diarrhea: Change at C3 D1: number analyzed (Participants) | 41 | 15
  Diarrhea: Change at C3 D1 | 7.32 (32.07) | 4.44 (30.52)
  Financial Difficulties: Change at C3 D1: number analyzed (Participants) | 40 | 15
  Financial Difficulties: Change at C3 D1 | 3.33 (24.81) | -2.22 (26.63)
  Global QoL: Change at C4 D1: number analyzed (Participants) | 30 | 12
  Global QoL: Change at C4 D1 | -6.67 (21.04) | -1.03 (15.27)
  Physical Functioning: Change at C4 D1: number analyzed (Participants) | 32 | 13
  Physical Functioning: Change at C4 D1 | -6.67 (23.15) | -1.03 (15.36)
  Role Functioning: Change at C4 D1: number analyzed (Participants) | 32 | 12
  Role Functioning: Change at C4 D1 | -7.81 (29.63) | 9.72 (36.56)
  Emotional Functioning: Change at C4 D1: number analyzed (Participants) | 31 | 12
  Emotional Functioning: Change at C4 D1 | -3.23 (22.64) | 9.03 (36.56)
  Cognitive Functioning: Change at C4 D1: number analyzed (Participants) | 31 | 12
  Cognitive Functioning: Change at C4 D1 | -6.99 (25.74) | 0.00 (15.89)
  Social Functioning: Change at C4 D1: number analyzed (Participants) | 31 | 11
  Social Functioning: Change at C4 D1 | -8.60 (35.45) | -1.52 (24.10)
  Fatigue: Change at C4 D1: number analyzed (Participants) | 32 | 13
  Fatigue: Change at C4 D1 | 7.47 (25.19) | -3.42 (25.41)
  Nausea and Vomiting: Change at C4 D1: number analyzed (Participants) | 32 | 13
  Nausea and Vomiting: Change at C4 D1 | -4.69 (19.96) | 6.41 (18.68)
  Pain: Change at C4 D1: number analyzed (Participants) | 32 | 13
  Pain: Change at C4 D1 | -16.67 (29.02) | -11.54 (28.37)
  Dyspnea: Change at C4 D1: number analyzed (Participants) | 31 | 13
  Dyspnea: Change at C4 D1 | 0.00 (28.54) | -5.13 (29.96)
  Insomnia: Change at C4 D1: number analyzed (Participants) | 32 | 13
  Insomnia: Change at C4 D1 | -11.46 (28.85) | -5.13 (32.90)
  Appetite loss: Change at C4 D1: number analyzed (Participants) | 32 | 12
  Appetite loss: Change at C4 D1 | 6.25 (36.35) | -2.78 (33.21)
  Constipation: Change at C4 D1: number analyzed (Participants) | 30 | 12
  Constipation: Change at C4 D1 | -24.44 (37.07) | -25.00 (40.51)
  Diarrhea: Change at C4 D1: number analyzed (Participants) | 31 | 12
  Diarrhea: Change at C4 D1 | 7.53 (39.17) | 5.56 (34.33)
  Financial Difficulties: Change at C4 D1: number analyzed (Participants) | 29 | 12
  Financial Difficulties: Change at C4 D1 | 1.15 (22.68) | -8.33 (20.72)
  Global QoL: Change at C5 D1: number analyzed (Participants) | 26 | 7
  Global QoL: Change at C5 D1 | -9.29 (27.82) | 10.71 (21.36)
  Physical Functioning: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Physical Functioning: Change at C5 D1 | -8.57 (23.08) | 0.00 (22.25)
  Role Functioning: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Role Functioning: Change at C5 D1 | -8.93 (29.22) | 7.14 (28.64)
  Emotional Functioning: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Emotional Functioning: Change at C5 D1 | -3.87 (22.96) | 20.24 (14.32)
  Cognitive Functioning: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Cognitive Functioning: Change at C5 D1 | -2.38 (24.73) | 7.14 (16.27)
  Social Functioning: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Social Functioning: Change at C5 D1 | -15.48 (33.92) | 4.76 (23.00)
  Fatigue: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Fatigue: Change at C5 D1 | 9.72 (28.59) | -15.28 (17.76)
  Nausea and Vomiting: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Nausea and Vomiting: Change at C5 D1 | 0.00 (26.06) | -6.25 (15.27)
  Pain: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Pain: Change at C5 D1 | -5.36 (34.26) | -25.00 (26.73)
  Dyspnea: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Dyspnea: Change at C5 D1 | 9.52 (27.00) | -12.50 (24.80)
  Insomnia: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Insomnia: Change at C5 D1 | -19.05 (35.63) | -29.17 (33.03)
  Appetite loss: Change at C5 D1: number analyzed (Participants) | 28 | 8
  Appetite loss: Change at C5 D1 | 0.00 (42.55) | -20.83 (43.42)
  Constipation: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Constipation: Change at C5 D1 | -21.43 (35.39) | -33.33 (38.49)
  Diarrhea: Change at C5 D1: number analyzed (Participants) | 28 | 7
  Diarrhea: Change at C5 D1 | 7.14 (33.16) | -4.76 (29.99)
  Financial Difficulties: Change at C5 D1: number analyzed (Participants) | 27 | 6
  Financial Difficulties: Change at C5 D1 | 0.00 (22.65) | 0.00 (36.51)
  Global QoL: Change at C6 D1: number analyzed (Participants) | 17 | 3
  Global QoL: Change at C6 D1 | -14.22 (20.36) | -5.56 (12.73)
  Physical Functioning: Change at C6 D1: number analyzed (Participants) | 19 | 2
  Physical Functioning: Change at C6 D1 | -6.32 (25.38) | 6.67 (18.86)
  Role Functioning: Change at C6 D1: number analyzed (Participants) | 19 | 2
  Role Functioning: Change at C6 D1 | -9.65 (27.95) | 16.67 (47.14)
  Emotional Functioning: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Emotional Functioning: Change at C6 D1 | 2.19 (15.92) | 8.33 (14.43)
  Cognitive Functioning: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Cognitive Functioning: Change at C6 D1 | -0.88 (18.82) | 11.11 (9.62)
  Social Functioning: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Social Functioning: Change at C6 D1 | -2.63 (27.92) | -16.67 (16.67)
  Fatigue: Change at C6 D1: number analyzed (Participants) | 19 | 2
  Fatigue: Change at C6 D1 | 6.73 (24.19) | -16.67 (39.28)
  Nausea and Vomiting: Change at C6 D1: number analyzed (Participants) | 19 | 2
  Nausea and Vomiting: Change at C6 D1 | -4.39 (22.80) | -8.33 (11.79)
  Pain: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Pain: Change at C6 D1 | -8.77 (30.11) | -33.33 (16.67)
  Dyspnea: Change at C6 D1(n=18,2): number analyzed (Participants) | 18 | 2
  Dyspnea: Change at C6 D1(n=18,2) | -1.85 (21.30) | 0.00 (47.14)
  Insomnia: Change at C6 D1: number analyzed (Participants) | 19 | 2
  Insomnia: Change at C6 D1 | -7.02 (30.59) | -16.67 (23.57)
  Appetite loss: Change at C6 D1(n=19,2): number analyzed (Participants) | 19 | 2
  Appetite loss: Change at C6 D1(n=19,2) | -3.51 (53.16) | -16.67 (70.71)
  Constipation: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Constipation: Change at C6 D1 | -10.53 (35.23) | -33.33 (33.33)
  Diarrhea: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Diarrhea: Change at C6 D1 | -1.75 (28.27) | 0.00 (33.33)
  Financial Difficulties: Change at C6 D1: number analyzed (Participants) | 19 | 3
  Financial Difficulties: Change at C6 D1 | 1.75 (13.49) | -22.22 (38.49)
  Global QoL: Change at C7 D1: number analyzed (Participants) | 9 | 3
  Global QoL: Change at C7 D1 | -4.63 (37.76) | -16.67 (14.43)
  Physical Functioning: Change at C7 D1: number analyzed (Participants) | 10 | 2
  Physical Functioning: Change at C7 D1 | -3.33 (24.80) | -22.22 (36.72)
  Role Functioning: Change at C7 D1: number analyzed (Participants) | 10 | 2
  Role Functioning: Change at C7 D1 | -15.00 (30.88) | 33.33 (70.71)
  Emotional Functioning: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Emotional Functioning: Change at C7 D1 | -8.33 (13.03) | -7.41 (21.58)
  Cognitive Functioning: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Cognitive Functioning: Change at C7 D1 | 1.67 (24.15) | -5.56 (9.62)
  Social Functioning: Change at C7 D1: number analyzed (Participants) | 10 | 2
  Social Functioning: Change at C7 D1 | -15.00 (41.16) | -25.00 (11.79)
  Fatigue: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Fatigue: Change at C7 D1 | -2.22 (25.01) | 14.81 (42.07)
  Nausea and Vomiting: Change at C7D1: number analyzed (Participants) | 10 | 3
  Nausea and Vomiting: Change at C7D1 | 1.67 (21.44) | 16.67 (0.00)
  Pain: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Pain: Change at C7 D1 | -3.33 (32.20) | -11.11 (41.94)
  Dyspnea: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Dyspnea: Change at C7 D1 | 16.67 (23.57) | 33.33 (33.33)
  Insomnia: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Insomnia: Change at C7 D1 | -10.00 (35.31) | 11.11 (38.49)
  Appetite loss: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Appetite loss: Change at C7 D1 | -10.00 (58.90) | 22.22 (50.92)
  Constipation: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Constipation: Change at C7 D1 | -13.33 (47.66) | -66.67 (57.74)
  Diarrhea: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Diarrhea: Change at C7 D1 | 3.33 (29.19) | 0.00 (0.00)
  Financial Difficulties: Change at C7 D1: number analyzed (Participants) | 10 | 3
  Financial Difficulties: Change at C7 D1 | -6.67 (21.08) | 0.00 (0.00)
  Global QoL: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Global QoL: Change at C8 D1 | -12.50 (33.62) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Physical Functioning Change at C8 D1: number analyzed (Participants) | 10 | 1
  Physical Functioning Change at C8 D1 | -10.67 (22.71) | -20.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Role Functioning: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Role Functioning: Change at C8 D1 | -13.33 (23.31) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Emotional Functioning: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Emotional Functioning: Change at C8 D1 | -7.50 (18.61) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cognitive Functioning: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Cognitive Functioning: Change at C8 D1 | 0.00 (22.22) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Social Functioning: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Social Functioning: Change at C8 D1 | -11.67 (34.29) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fatigue: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Fatigue: Change at C8 D1 | 4.44 (25.23) | 2.22 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Nausea and Vomiting: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Nausea and Vomiting: Change at C8 D1 | 0.00 (19.25) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pain: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Pain: Change at C8 D1 | -8.33 (37.06) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Dyspnea: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Dyspnea: Change at C8 D1 | 14.81 (29.40) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Insomnia: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Insomnia: Change at C8 D1 | -20.00 (47.66) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Appetite loss: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Appetite loss: Change at C8 D1 | -3.33 (48.30) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Constipation: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Constipation: Change at C8 D1 | -3.33 (29.19) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Diarrhea: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Diarrhea: Change at C8 D1 | 6.67 (37.84) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Financial Difficulties: Change at C8 D1: number analyzed (Participants) | 10 | 1
  Financial Difficulties: Change at C8 D1 | -3.33 (18.92) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Global QoL: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Global QoL: Change at C9 D1 | -17.71 (36.03) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Physical Functioning: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Physical Functioning: Change at C9 D1 | -6.67 (20.16) | -40.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Role Functioning: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Role Functioning: Change at C9 D1 | -29.17 (24.80) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Emotional Functioning: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Emotional Functioning: Change at C9 D1 | -3.13 (13.32) | -8.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cognitive Functioning: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Cognitive Functioning: Change at C9 D1 | -2.08 (28.78) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Social Functioning: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Social Functioning: Change at C9 D1 | -6.25 (47.09) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fatigue: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Fatigue: Change at C9 D1 | 18.06 (33.56) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Nausea and Vomiting: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Nausea and Vomiting: Change at C9 D1 | -8.33 (17.82) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pain: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Pain: Change at C9 D1 | 0.00 (30.86) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Dyspnea: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Dyspnea: Change at C9 D1 | 19.05 (26.23) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Insomnia: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Insomnia: Change at C9 D1 | -4.17 (33.03) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Appetite loss: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Appetite loss: Change at C9 D1 | 8.33 (63.62) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Constipation: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Constipation: Change at C9 D1 | -8.33 (38.83) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Diarrhea: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Diarrhea: Change at C9 D1 | 12.50 (43.42) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Financial Difficulties: Change at C9 D1: number analyzed (Participants) | 8 | 1
  Financial Difficulties: Change at C9 D1 | -4.17 (21.36) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Global QoL: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Global QoL: Change at C10 D1 | -16.67 (21.52) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Physical Functioning: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Physical Functioning: Change at C10 D1 | -19.05 (13.01) | -46.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Role Functioning: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Role Functioning: Change at C10 D1 | -23.81 (21.21) | -50.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Emotional Functioning: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Emotional Functioning: Change at C10 D1 | -20.24 (23.00) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cognitive Functioning: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Cognitive Functioning: Change at C10 D1 | -9.52 (21.21) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Social Functioning: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Social Functioning: Change at C10 D1 | -21.43 (31.50) | -50.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fatigue: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Fatigue: Change at C10 D1 | 25.40 (24.61) | 55.56 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Nausea and Vomiting: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Nausea and Vomiting: Change at C10 D1 | 0.00 (25.46) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pain: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Pain: Change at C10 D1 | 11.90 (35.63) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Dyspnea: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Dyspnea: Change at C10 D1 | 22.22 (27.22) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Insomnia: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Insomnia: Change at C10 D1 | 4.76 (23.00) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Appetite loss: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Appetite loss: Change at C10 D1 | 23.81 (46.00) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Constipation: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Constipation: Change at C10 D1 | -19.05 (37.80) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Diarrhea: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Diarrhea: Change at C10 D1 | 9.52 (31.71) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Financial Difficulties: Change at C10 D1: number analyzed (Participants) | 7 | 1
  Financial Difficulties: Change at C10 D1 | -4.76 (23.00) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Global QoL: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Global QoL: Change at C11 D1 | -38.89 (53.58) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Physical Functioning: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Physical Functioning: Change at C11 D1 | -24.44 (36.72) | -40.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Role Functioning: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Role Functioning: Change at C11 D1 | -38.89 (53.58) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Emotional Functioning: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Emotional Functioning: Change at C11 D1 | -25.00 (52.04) | -8.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cognitive Functioning: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Cognitive Functioning: Change at C11 D1 | -27.78 (63.10) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Social Functioning: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Social Functioning: Change at C11 D1 | -38.89 (53.58) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fatigue: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Fatigue: Change at C11 D1 | 37.04 (46.26) | 22.22 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Nausea and Vomiting: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Nausea and Vomiting: Change at C11 D1 | 27.78 (63.10) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pain: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Pain: Change at C11 D1 | 22.22 (69.39) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Dyspnea: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Dyspnea: Change at C11 D1 | 22.22 (69.39) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Insomnia: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Insomnia: Change at C11 D1 | 22.22 (69.39) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Appetite loss: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Appetite loss: Change at C11 D1 | 44.44 (50.92) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Constipation: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Constipation: Change at C11 D1 | 0.00 (33.33) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Diarrhea: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Diarrhea: Change at C11 D1 | 11.11 (19.25) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Financial Difficulties: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Financial Difficulties: Change at C11 D1 | -11.11 (19.25) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Global QoL: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Global QoL: Change at C12 D1 | -11.11 (17.35) |
  Physical Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Physical Functioning: Change at C12 D1 | -6.67 (6.67) |
  Role Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Role Functioning: Change at C12 D1 | -11.11 (19.25) |
  Emotional Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Emotional Functioning: Change at C12 D1 | -2.78 (20.97) |
  Cognitive Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Cognitive Functioning: Change at C12 D1 | 0.00 (16.67) |
  Social Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Social Functioning: Change at C12 D1 | -5.56 (9.62) |
  Fatigue: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Fatigue: Change at C12 D1 | 7.41 (12.83) |
  Nausea and Vomiting: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Nausea and Vomiting: Change at C12 D1 | 16.67 (60.09) |
  Pain: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Pain: Change at C12 D1 | -5.56 (9.62) |
  Dyspnea: Change at C12 D1: number analyzed (Participants) | 2 | 0
  Dyspnea: Change at C12 D1 | 0.00 (0.00) |
  Insomnia: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Insomnia: Change at C12 D1 | -11.11 (19.25) |
  Appetite loss: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Appetite loss: Change at C12 D1 | 22.22 (19.25) |
  Constipation: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Constipation: Change at C12 D1 | -22.22 (38.49) |
  Diarrhea: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Diarrhea: Change at C12 D1 | 22.22 (19.25) |
  Financial Difficulties: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Financial Difficulties: Change at C12 D1 | -11.11 (19.25) |
  Global QoL: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Global QoL: Change at C13 D1 | -50.00 (35.36) |
  Physical Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Physical Functioning: Change at C13 D1 | -23.33 (33.00) |
  Role Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Role Functioning: Change at C13 D1 | -41.67 (35.36) |
  Emotional Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Emotional Functioning: Change at C13 D1 | -8.33 (11.79) |
  Cognitive Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Cognitive Functioning: Change at C13 D1 | 0.00 (0.00) |
  Social Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Social Functioning: Change at C13 D1 | -8.33 (35.36) |
  Fatigue: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Fatigue: Change at C13 D1 | 33.33 (47.14) |
  Nausea and Vomiting: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Nausea and Vomiting: Change at C13 D1 | -8.33 (35.36) |
  Pain: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Pain: Change at C13 D1 | 41.67 (58.93) |
  Dyspnea: Change at C13 D1: number analyzed (Participants) | 1 | 0
  Dyspnea: Change at C13 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Insomnia: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Insomnia: Change at C13 D1 | 0.00 (0.00) |
  Appetite loss: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Appetite loss: Change at C13 D1 | 33.33 (47.14) |
  Constipation: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Constipation: Change at C13 D1 | -16.67 (23.57) |
  Diarrhea: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Diarrhea: Change at C13 D1 | 16.67 (23.57) |
  Financial Difficulties: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Financial Difficulties: Change at C13 D1 | -16.67 (23.57) |
  Global QoL: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Global QoL: Change at C14 D1 | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Physical Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Physical Functioning: Change at C14 D1 | -6.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Role Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Role Functioning: Change at C14 D1 | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Emotional Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Emotional Functioning: Change at C14 D1 | -8.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Cognitive Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Cognitive Functioning: Change at C14 D1 | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Social Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Social Functioning: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Fatigue: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Fatigue: Change at C14 D1 | 22.22 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Nausea and Vomiting: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Nausea and Vomiting: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Pain: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Pain: Change at C14 D1 | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Dyspnea: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Dyspnea: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Insomnia: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Insomnia: Change at C14 D1 | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Appetite loss: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Appetite loss: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Constipation: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Constipation: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Diarrhea: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Diarrhea: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Financial Difficulties: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Financial Difficulties: Change at C14 D1 | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Global QoL: Change at EoS: number analyzed (Participants) | 2 | 1
  Global QoL: Change at EoS | -54.17 (29.46) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Physical Functioning: Change at EoS: number analyzed (Participants) | 2 | 1
  Physical Functioning: Change at EoS | -70.00 (4.71) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Role Functioning: Change at EoS: number analyzed (Participants) | 2 | 1
  Role Functioning: Change at EoS | -33.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Emotional Functioning: Change at EoS: number analyzed (Participants) | 2 | 1
  Emotional Functioning: Change at EoS | -66.67 (35.36) | -25.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cognitive Functioning: Change at EoS: number analyzed (Participants) | 2 | 1
  Cognitive Functioning: Change at EoS | -66.67 (0.00) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Social Functioning: Change at EoS: number analyzed (Participants) | 2 | 1
  Social Functioning: Change at EoS | -83.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fatigue: Change at EoS: number analyzed (Participants) | 2 | 1
  Fatigue: Change at EoS | 55.56 (15.71) | -11.11 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Nausea and Vomiting: Change at EoS: number analyzed (Participants) | 2 | 1
  Nausea and Vomiting: Change at EoS | 33.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pain: Change at EoS: number analyzed (Participants) | 2 | 1
  Pain: Change at EoS | 41.67 (82.50) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Dyspnea: Change at EoS: number analyzed (Participants) | 2 | 1
  Dyspnea: Change at EoS | 83.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Insomnia: Change at EoS: number analyzed (Participants) | 2 | 1
  Insomnia: Change at EoS | 66.67 (47.14) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Appetite loss: Change at EoS: number analyzed (Participants) | 2 | 1
  Appetite loss: Change at EoS | 50.00 (70.71) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Constipation: Change at EoS: number analyzed (Participants) | 2 | 1
  Constipation: Change at EoS | -16.67 (117.85) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Diarrhea: Change at EoS: number analyzed (Participants) | 2 | 1
  Diarrhea: Change at EoS | 33.33 (47.14) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Financial Difficulties: Change at EoS: number analyzed (Participants) | 2 | 1
  Financial Difficulties: Change at EoS | -16.67 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -8.44, 95% CI 2-sided [-19.06 to 2.19]
Statistical Analysis 2: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.02, 95% CI 2-sided [-15.4 to 3.36]
Statistical Analysis 3: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -9.32, 95% CI 2-sided [-23.77 to 5.12]
Statistical Analysis 4: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.73, 95% CI 2-sided [-15.25 to 5.79]
Statistical Analysis 5: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -5.11, 95% CI 2-sided [-15.83 to 5.61]
Statistical Analysis 6: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-18.72 to 12.06]
Statistical Analysis 7: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.41, 95% CI 2-sided [-1.62 to 22.44]
Statistical Analysis 8: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.30, 95% CI 2-sided [-16.55 to 7.96]
Statistical Analysis 9: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 7.37, 95% CI 2-sided [-7.57 to 22.32]
Statistical Analysis 10: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.51, 95% CI 2-sided [-1.28 to 26.30]
Statistical Analysis 11: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.90, 95% CI 2-sided [-5.70 to 25.49]
Statistical Analysis 12: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.63, 95% CI 2-sided [-4.81 to 32.07]
Statistical Analysis 13: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 4.67, 95% CI 2-sided [-11.62 to 20.96]
Statistical Analysis 14: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-15.1 to 12.54]
Statistical Analysis 15: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.43, 95% CI 2-sided [-4.67 to 15.53]
Statistical Analysis 16: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -15.83, 95% CI 2-sided [-32.34 to 0.67]
Statistical Analysis 17: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.58, 95% CI 2-sided [-24.12 to 0.96]
Statistical Analysis 18: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -18.65, 95% CI 2-sided [-35.47 to -1.83]
Statistical Analysis 19: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -13.92, 95% CI 2-sided [-29.16 to 1.32]
Statistical Analysis 20: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.10, 95% CI 2-sided [-20.97 to 6.77]
Statistical Analysis 21: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -9.62, 95% CI 2-sided [-28.28 to 9.04]
Statistical Analysis 22: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.14, 95% CI 2-sided [-1.27 to 33.54]
Statistical Analysis 23: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-18.78 to 15.18]
Statistical Analysis 24: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.59, 95% CI 2-sided [-3.22 to 36.39]
Statistical Analysis 25: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.39, 95% CI 2-sided [-5.68 to 26.47]
Statistical Analysis 26: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-20.19 to 23.36]
Statistical Analysis 27: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.24, 95% CI 2-sided [-7.62 to 40.1]
Statistical Analysis 28: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 2.76, 95% CI 2-sided [-17.49 to 23.02]
Statistical Analysis 29: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 2.87, 95% CI 2-sided [-16.29 to 22.03]
Statistical Analysis 30: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [-9.81 to 20.92]
Statistical Analysis 31: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -5.97, 95% CI 2-sided [-19.52 to 7.57]
Statistical Analysis 32: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -5.64, 95% CI 2-sided [-19.75 to 8.46]
Statistical Analysis 33: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -17.53, 95% CI 2-sided [-39.11 to 4.05]
Statistical Analysis 34: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -12.25, 95% CI 2-sided [-26.5 to 2.00]
Statistical Analysis 35: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.99, 95% CI 2-sided [-23.13 to 9.15]
Statistical Analysis 36: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.09, 95% CI 2-sided [-30.48 to 16.31]
Statistical Analysis 37: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.88, 95% CI 2-sided [-5.86 to 27.63]
Statistical Analysis 38: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.10, 95% CI 2-sided [-24.11 to 1.91]
Statistical Analysis 39: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -5.13, 95% CI 2-sided [-24.26 to 14.00]
Statistical Analysis 40: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.13, 95% CI 2-sided [-14.18 to 24.44]
Statistical Analysis 41: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.33, 95% CI 2-sided [-26.25 to 13.59]
Statistical Analysis 42: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.03, 95% CI 2-sided [-15.26 to 33.32]
Statistical Analysis 43: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-25.71 to 26.82]
Statistical Analysis 44: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [-24.07 to 28.01]
Statistical Analysis 45: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.48, 95% CI 2-sided [-5.89 to 24.86]
Statistical Analysis 46: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -20.01, 95% CI 2-sided [-43.19 to 3.17]
Statistical Analysis 47: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -8.57, 95% CI 2-sided [-27.24 to 10.10]
Statistical Analysis 48: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.07, 95% CI 2-sided [-41.10 to 8.96]
Statistical Analysis 49: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -24.11, 95% CI 2-sided [-42.72 to -5.50]
Statistical Analysis 50: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -9.52, 95% CI 2-sided [-29.66 to 10.61]
Statistical Analysis 51: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -20.24, 95% CI 2-sided [-47.93 to 7.46]
Statistical Analysis 52: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [3.23 to 46.77]
Statistical Analysis 53: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 6.25, 95% CI 2-sided [-13.49 to 25.99]
Statistical Analysis 54: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 19.64, 95% CI 2-sided [-7.12 to 46.41]
Statistical Analysis 55: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.02, 95% CI 2-sided [0.38 to 43.66]
Statistical Analysis 56: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.12, 95% CI 2-sided [-18.49 to 38.73]
Statistical Analysis 57: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.83, 95% CI 2-sided [-13.98 to 55.65]
Statistical Analysis 58: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.90, 95% CI 2-sided [-19.02 to 42.83]
Statistical Analysis 59: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.90, 95% CI 2-sided [-16.13 to 39.94]
Statistical Analysis 60: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-23.38 to 23.38]
Statistical Analysis 61: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -8.66, 95% CI 2-sided [-34.53 to 17.21]
Statistical Analysis 62: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -12.98, 95% CI 2-sided [-52.01 to 26.04]
Statistical Analysis 63: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -26.32, 95% CI 2-sided [-71.87 to 19.24]
Statistical Analysis 64: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.14, 95% CI 2-sided [-26.59 to 14.31]
Statistical Analysis 65: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.99, 95% CI 2-sided [-35.46 to 11.48]
Statistical Analysis 66: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.04, 95% CI 2-sided [-20.97 to 49.04]
Statistical Analysis 67: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.39, 95% CI 2-sided [-15.83 to 62.61]
Statistical Analysis 68: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [-30.84 to 38.73]
Statistical Analysis 69: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 24.56, 95% CI 2-sided [-13.08 to 62.20]
Statistical Analysis 70: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-38.65 to 34.94]
Statistical Analysis 71: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.65, 95% CI 2-sided [-37.43 to 56.73]
Statistical Analysis 72: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.16, 95% CI 2-sided [-71.22 to 97.54]
Statistical Analysis 73: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.81, 95% CI 2-sided [-22.61 to 68.22]
Statistical Analysis 74: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-39.10 to 35.59]
Statistical Analysis 75: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.98, 95% CI 2-sided [1.09 to 46.86]
Statistical Analysis 76: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.04, 95% CI 2-sided [-39.03 to 63.11]
Statistical Analysis 77: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 18.89, 95% CI 2-sided [-20.74 to 58.52]
Statistical Analysis 78: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -48.33, 95% CI 2-sided [-111.94 to 15.28]
Statistical Analysis 79: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-22.59 to 20.74]
Statistical Analysis 80: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 7.22, 95% CI 2-sided [-24.98 to 39.43]
Statistical Analysis 81: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.00, 95% CI 2-sided [-57.71 to 77.71]
Statistical Analysis 82: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -17.04, 95% CI 2-sided [-58.87 to 24.79]
Statistical Analysis 83: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -15.00, 95% CI 2-sided [-43.10 to 13.10]
Statistical Analysis 84: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 7.78, 95% CI 2-sided [-41.75 to 57.30]
Statistical Analysis 85: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-53.79 to 20.46]
Statistical Analysis 86: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -21.11, 95% CI 2-sided [-73.14 to 30.92]
Statistical Analysis 87: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -32.22, 95% CI 2-sided [-115.58 to 51.13]
Statistical Analysis 88: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 53.33, 95% CI 2-sided [-18.60 to 125.26]
Statistical Analysis 89: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.33, 95% CI 2-sided [-34.92 to 41.58]
Statistical Analysis 90: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.67, 95% CI 2-sided [-34.3 to 20.96]
Statistical Analysis 91: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.83, 95% CI 2-sided [-58.94 to 100.60]
Statistical Analysis 92: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.33, 95% CI 2-sided [-44.54 to 63.20]
Statistical Analysis 93: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.00, 95% CI 2-sided [-35.30 to 75.30]
Statistical Analysis 94: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.50, 95% CI 2-sided [-51.66 to 36.66]
Statistical Analysis 95: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.67, 95% CI 2-sided [-36.06 to 69.39]
Statistical Analysis 96: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.00, 95% CI 2-sided [-76.36 to 86.36]
Statistical Analysis 97: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -17.78, 95% CI 2-sided [-77.63 to 42.08]
Statistical Analysis 98: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-62.33 to 28.99]
Statistical Analysis 99: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 8.33, 95% CI 2-sided [-79.59 to 96.26]
Statistical Analysis 100: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -18.52, 95% CI 2-sided [-89.98 to 52.94]
Statistical Analysis 101: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -20.00, 95% CI 2-sided [-133.08 to 93.08]
Statistical Analysis 102: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -36.67, 95% CI 2-sided [-151.27 to 77.94]
Statistical Analysis 103: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-72.58 to 65.91]
Statistical Analysis 104: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 73.33, 95% CI 2-sided [-16.45 to 163.12]
Statistical Analysis 105: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-48.23 to 41.56]
Statistical Analysis 106: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.62, 95% CI 2-sided [-74.75 to 106.00]
Statistical Analysis 107: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 33.33, 95% CI 2-sided [-17.22 to 83.89]
Statistical Analysis 108: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 4.17, 95% CI 2-sided [-58.04 to 66.37]
Statistical Analysis 109: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.21, 95% CI 2-sided [-28.19 to 38.61]
Statistical Analysis 110: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 31.25, 95% CI 2-sided [-40.94 to 103.44]
Statistical Analysis 111: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.08, 95% CI 2-sided [-91.02 to 145.18]
Statistical Analysis 112: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -15.28, 95% CI 2-sided [-99.46 to 68.90]
Statistical Analysis 113: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -25.00, 95% CI 2-sided [-69.69 to 19.69]
Statistical Analysis 114: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-77.40 to 77.40]
Statistical Analysis 115: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -14.29, 95% CI 2-sided [-82.89 to 54.32]
Statistical Analysis 116: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.17, 95% CI 2-sided [-87.02 to 78.69]
Statistical Analysis 117: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -25.00, 95% CI 2-sided [-184.57 to 134.57]
Statistical Analysis 118: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -8.33, 95% CI 2-sided [-105.73 to 89.06]
Statistical Analysis 119: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 79.17, 95% CI 2-sided [-29.72 to 188.06]
Statistical Analysis 120: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.17, 95% CI 2-sided [-57.74 to 49.41]
Statistical Analysis 121: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.67, 95% CI 2-sided [-39.62 to 72.95]
Statistical Analysis 122: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.62, 95% CI 2-sided [-6.42 to 61.66]
Statistical Analysis 123: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 26.19, 95% CI 2-sided [-29.28 to 81.66]
Statistical Analysis 124: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.57, 95% CI 2-sided [-63.74 to 56.6]
Statistical Analysis 125: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.81, 95% CI 2-sided [-31.66 to 79.28]
Statistical Analysis 126: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 28.57, 95% CI 2-sided [-53.82 to 110.96]
Statistical Analysis 127: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -30.16, 95% CI 2-sided [-94.53 to 34.21]
Statistical Analysis 128: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-83.26 to 49.93]
Statistical Analysis 129: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.76, 95% CI 2-sided [-97.98 to 88.45]
Statistical Analysis 130: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.11, 95% CI 2-sided [-86.68 to 64.46]
Statistical Analysis 131: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 4.76, 95% CI 2-sided [-55.41 to 64.93]
Statistical Analysis 132: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -9.52, 95% CI 2-sided [-129.86 to 110.82]
Statistical Analysis 133: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -19.05, 95% CI 2-sided [-117.92 to 79.82]
Statistical Analysis 134: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 76.19, 95% CI 2-sided [-6.75 to 159.13]
Statistical Analysis 135: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.76, 95% CI 2-sided [-64.93 to 55.41]
Statistical Analysis 136: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -5.56, 95% CI 2-sided [-271.74 to 260.62]
Statistical Analysis 137: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.56, 95% CI 2-sided [-166.87 to 197.98]
Statistical Analysis 138: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.78, 95% CI 2-sided [-238.4 to 293.96]
Statistical Analysis 139: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-275.22 to 241.89]
Statistical Analysis 140: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [-307.94 to 319.05]
Statistical Analysis 141: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.78, 95% CI 2-sided [-238.40 to 293.96]
Statistical Analysis 142: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.81, 95% CI 2-sided [-215.01 to 244.64]
Statistical Analysis 143: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.11, 95% CI 2-sided [-302.38 to 324.60]
Statistical Analysis 144: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 38.89, 95% CI 2-sided [-305.85 to 383.63]
Statistical Analysis 145: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.11, 95% CI 2-sided [-355.85 to 333.63]
Statistical Analysis 146: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.22, 95% CI 2-sided [-322.52 to 366.97]
Statistical Analysis 147: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 44.44, 95% CI 2-sided [-208.53 to 297.42]
Statistical Analysis 148: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-165.61 to 165.61]
Statistical Analysis 149: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 77.78, 95% CI 2-sided [-17.84 to 173.39]
Statistical Analysis 150: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.11, 95% CI 2-sided [-106.73 to 84.5]
Statistical Analysis 151: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in global QoL at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -54.17, 95% CI 2-sided [-512.66 to 404.33]
Statistical Analysis 152: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in physical functioning at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -70.00, 95% CI 2-sided [-143.36 to 3.36]
Statistical Analysis 153: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in role functioning at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -33.33, 95% CI 2-sided [-400.13 to 333.46]
Statistical Analysis 154: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in emotional functioning at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -41.67, 95% CI 2-sided [-591.86 to 508.53]
Statistical Analysis 155: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cognitive functioning at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -66.67, 95% CI 2-sided [-66.67 to -66.67]
Statistical Analysis 156: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in social functioning at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -83.33, 95% CI 2-sided [-450.13 to 283.46]
Statistical Analysis 157: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fatigue at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 66.67, 95% CI 2-sided [-177.86 to 311.2]
Statistical Analysis 158: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in nausea and vomiting at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 33.33, 95% CI 2-sided [-333.46 to 400.13]
Statistical Analysis 159: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pain at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [-1258.79 to 1308.79]
Statistical Analysis 160: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in dyspnea at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 83.33, 95% CI 2-sided [-283.46 to 450.13]
Statistical Analysis 161: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in insomnia at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 33.33, 95% CI 2-sided [-700.26 to 766.93]
Statistical Analysis 162: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in appetite loss at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 50.00, 95% CI 2-sided [-1050.39 to 1150.39]
Statistical Analysis 163: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in constipation at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-1850.65 to 1817.32]
Statistical Analysis 164: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in diarrhea at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 33.33, 95% CI 2-sided [-700.26 to 766.93]
Statistical Analysis 165: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in financial difficulties at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -16.67, 95% CI 2-sided [-383.46 to 350.13]

17. Secondary Outcome: Change From Baseline in 26-item Pancreatic Cancer-specific Quality of Life Questionnaire (QLQ-PAN26) Score at Day 1 of Every Cycle and End of Study
Description: QLQ-PAN26 consists of 26 questions (Qs) relating to disease symptoms, treatment (Tx) side effects and emotional issues specific to pancreatic cancer (PC). Questions include on altered bowel habits, pain, dietary changes, disease and Tx-related symptoms and issues related to the emotional and social well-being of participants with PC. All 26 Qs are answered on 4-point Likert scale ranging from '1=not at all' to 4='very much' and subsequently transformed into scales that range from 0-100. Higher scores on functioning scales=better functioning; higher scores on the symptom scales=more symptoms.
Time Frame: Phase 2 baseline [Day (D) 1 of Cycle (C)1], Day 1 of all subsequent cycles up to Cycle 14 and end of study (EoS).
Population: Phase 2 ITT population was the primary analysis population. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. n signifies the number of participants evaluable for the respective scale at the respective time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Axitinib + Gemcitabine | Gemcitabine
Number analyzed (Participants) | 59 | 27
units on a scale
  Pancreatic Pain: Baseline | 37.52 (27.88) | 38.89 (21.18)
  Eating Related Items: Baseline | 40.40 (35.18) | 33.95 (27.92)
  Altered Bowel Habits: Baseline | 22.32 (26.19) | 25.31 (28.26)
  Jaundice: Baseline: number analyzed (Participants) | 59 | 26
  Jaundice: Baseline | 9.89 (18.34) | 15.38 (23.06)
  Body Image: Baseline | 31.64 (29.80) | 26.54 (25.84)
  Health Care Satisfaction: Baseline | 79.38 (27.57) | 69.75 (25.33)
  Sexual Functioning: Baseline: number analyzed (Participants) | 56 | 23
  Sexual Functioning: Baseline | 44.35 (34.42) | 57.97 (37.56)
  Ascites: Baseline | 37.29 (31.00) | 25.93 (25.04)
  Indigestion: Baseline | 24.86 (28.09) | 30.86 (34.50)
  Flatulence: Baseline | 35.59 (32.67) | 39.51 (29.29)
  Cachexia: Baseline | 33.62 (25.43) | 31.48 (23.72)
  Side Effects: Baseline: number analyzed (Participants) | 59 | 26
  Side Effects: Baseline | 27.78 (24.80) | 27.35 (21.77)
  Fear of Future Health: Baseline: number analyzed (Participants) | 58 | 27
  Fear of Future Health: Baseline | 63.22 (31.03) | 59.26 (33.76)
  Ability to Plan Future: Baseline | 39.55 (35.27) | 41.98 (36.51)
  Pancreatic Pain: Change at C2 D1: number analyzed (Participants) | 44 | 22
  Pancreatic Pain: Change at C2 D1 | -11.05 (25.39) | -13.64 (22.05)
  Eating Related Items: Change at C2 D1: number analyzed (Participants) | 44 | 22
  Eating Related Items: Change at C2 D1 | -0.38 (34.19) | -3.79 (27.67)
  Altered Bowel Habits: Change at C2 D1: number analyzed (Participants) | 44 | 22
  Altered Bowel Habits: Change at C2 D1 | 8.33 (28.19) | -11.36 (22.05)
  Jaundice: Change at C2 D1: number analyzed (Participants) | 44 | 21
  Jaundice: Change at C2 D1 | 0.00 (20.65) | -12.70 (25.22)
  Body Image: Change at C2 D1: number analyzed (Participants) | 44 | 21
  Body Image: Change at C2 D1 | 7.95 (26.53) | -7.14 (25.04)
  Health Care Satisfaction: Change at C2 D1: number analyzed (Participants) | 43 | 21
  Health Care Satisfaction: Change at C2 D1 | 0.39 (34.60) | -3.97 (37.60)
  Sexual Functioning: Change at C2 D1: number analyzed (Participants) | 39 | 17
  Sexual Functioning: Change at C2 D1 | -2.56 (22.14) | 18.63 (38.59)
  Ascites: Change at C2 D1: number analyzed (Participants) | 43 | 22
  Ascites: Change at C2 D1 | -10.85 (36.89) | -3.03 (22.79)
  Indigestion: Change at C2 D1: number analyzed (Participants) | 43 | 22
  Indigestion: Change at C2 D1 | -4.65 (24.75) | -10.61 (37.64)
  Flatulence: Change at C2 D1: number analyzed (Participants) | 44 | 22
  Flatulence: Change at C2 D1 | 5.30 (34.43) | -9.09 (21.04)
  Cachexia: Change at C2 D1: number analyzed (Participants) | 44 | 22
  Cachexia: Change at C2 D1 | 9.47 (19.15) | -3.03 (17.55)
  Side Effects: Change at C2 D1: number analyzed (Participants) | 44 | 21
  Side Effects: Change at C2 D1 | 7.70 (16.39) | -3.17 (20.90)
  Fear of Future Health: Change at C2 D1: number analyzed (Participants) | 43 | 21
  Fear of Future Health: Change at C2 D1 | -2.33 (23.45) | 0.00 (31.62)
  Ability to Plan Future: Change at C2 D1: number analyzed (Participants) | 44 | 20
  Ability to Plan Future: Change at C2 D1 | 4.55 (35.65) | -1.67 (27.52)
  Pancreatic Pain: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Pancreatic Pain: Change at C3 D1 | -8.92 (24.62) | -23.78 (20.61)
  Eating Related Items: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Eating Related Items: Change at C3 D1 | 3.07 (37.34) | -10.42 (28.46)
  Altered Bowel Habits: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Altered Bowel Habits: Change at C3 D1 | 10.53 (31.34) | -8.33 (31.03)
  Jaundice: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Jaundice: Change at C3 D1 | 2.19 (13.52) | -9.38 (26.51)
  Body Image: Change at C3 D1: number analyzed (Participants) | 37 | 16
  Body Image: Change at C3 D1 | 13.51 (30.89) | -5.21 (29.01)
  Health Care Satisfaction: Change at C3 D1: number analyzed (Participants) | 37 | 16
  Health Care Satisfaction: Change at C3 D1 | -5.41 (40.07) | 5.21 (24.88)
  Sexual Functioning: Change at C3 D1: number analyzed (Participants) | 32 | 15
  Sexual Functioning: Change at C3 D1 | -3.13 (21.77) | -4.44 (31.79)
  Ascites: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Ascites: Change at C3 D1 | -2.63 (28.35) | -4.17 (23.96)
  Indigestion: Change at C3 D1: number analyzed (Participants) | 37 | 15
  Indigestion: Change at C3 D1 | -4.50 (34.39) | -15.56 (37.52)
  Flatulence: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Flatulence: Change at C3 D1 | 9.65 (37.09) | 6.25 (27.81)
  Cachexia: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Cachexia: Change at C3 D1 | 14.47 (24.56) | 5.21 (17.97)
  Side Effects: Change at C3 D1: number analyzed (Participants) | 38 | 16
  Side Effects: Change at C3 D1 | 11.55 (27.41) | -7.64 (26.28)
  Fear of Future Health: Change at C3 D1: number analyzed (Participants) | 35 | 15
  Fear of Future Health: Change at C3 D1 | -2.86 (34.65) | -2.22 (42.66)
  Ability to Plan Future: Change at C3 D1: number analyzed (Participants) | 37 | 16
  Ability to Plan Future: Change at C3 D1 | 9.01 (43.50) | -12.50 (34.16)
  Pancreatic Pain: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Pancreatic Pain: Change at C4 D1 | -18.30 (26.90) | -14.10 (22.92)
  Eating Related Items: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Eating Related Items: Change at C4 D1 | -7.47 (26.57) | 5.13 (36.88)
  Altered Bowel Habits: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Altered Bowel Habits: Change at C4 D1 | 16.09 (35.21) | 3.85 (28.99)
  Jaundice: Change at C4 D1: number analyzed (Participants) | 29 | 12
  Jaundice: Change at C4 D1 | 1.72 (19.59) | -11.11 (16.41)
  Body Image: Change at C4 D1: number analyzed (Participants) | 26 | 13
  Body Image: Change at C4 D1 | 12.82 (31.02) | 8.97 (26.01)
  Health Care Satisfaction: Change at C4 D1: number analyzed (Participants) | 26 | 13
  Health Care Satisfaction: Change at C4 D1 | -1.92 (49.51) | -8.97 (29.36)
  Sexual Functioning: Change at C4 D1: number analyzed (Participants) | 22 | 12
  Sexual Functioning: Change at C4 D1 | -5.30 (27.88) | -2.78 (40.72)
  Ascites: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Ascites: Change at C4 D1 | -6.90 (25.79) | 2.56 (28.74)
  Indigestion: Change at C4 D1: number analyzed (Participants) | 28 | 13
  Indigestion: Change at C4 D1 | -9.52 (33.77) | -2.56 (37.17)
  Flatulence: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Flatulence: Change at C4 D1 | 1.15 (39.32) | -2.56 (25.32)
  Cachexia: Change at C4 D1: number analyzed (Participants) | 29 | 13
  Cachexia: Change at C4 D1 | 9.20 (29.07) | -3.85 (24.68)
  Side Effects: Change at C4 D1: number analyzed (Participants) | 29 | 12
  Side Effects: Change at C4 D1 | 11.88 (28.59) | -3.24 (19.88)
  Fear of Future Health: Change at C4 D1: number analyzed (Participants) | 24 | 13
  Fear of Future Health: Change at C4 D1 | -2.78 (41.61) | 5.13 (38.12)
  Ability to Plan Future: Change at C4 D1: number analyzed (Participants) | 26 | 13
  Ability to Plan Future: Change at C4 D1 | 10.26 (53.97) | -5.13 (46.84)
  Pancreatic Pain: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Pancreatic Pain: Change at C5 D1 | -7.26 (27.99) | -18.52 (24.22)
  Eating Related Items: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Eating Related Items: Change at C5 D1 | 0.00 (45.22) | -7.41 (26.50)
  Altered Bowel Habits: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Altered Bowel Habits: Change at C5 D1 | 13.46 (30.92) | -14.81 (29.40)
  Jaundice: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Jaundice: Change at C5 D1 | 3.85 (19.04) | -20.37 (36.11)
  Body Image: Change at C5 D1: number analyzed (Participants) | 25 | 9
  Body Image: Change at C5 D1 | 14.00 (28.74) | -11.11 (39.97)
  Health Care Satisfaction: Change at C5 D1: number analyzed (Participants) | 25 | 9
  Health Care Satisfaction: Change at C5 D1 | -2.67 (51.52) | 7.41 (34.47)
  Sexual Functioning: Change at C5 D1: number analyzed (Participants) | 19 | 9
  Sexual Functioning: Change at C5 D1 | -1.75 (20.71) | 1.85 (24.22)
  Ascites: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Ascites: Change at C5 D1 | -5.13 (24.39) | -11.11 (40.82)
  Indigestion: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Indigestion: Change at C5 D1 | -3.85 (28.79) | -25.93 (49.38)
  Flatulence: Change at C5 D1: number analyzed (Participants) | 25 | 9
  Flatulence: Change at C5 D1 | -1.33 (28.02) | -11.11 (40.82)
  Cachexia: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Cachexia: Change at C5 D1 | 10.26 (36.84) | -5.56 (18.63)
  Side Effects: Change at C5 D1: number analyzed (Participants) | 26 | 9
  Side Effects: Change at C5 D1 | 10.04 (28.55) | -11.73 (17.22)
  Fear of Future Health: Change at C5 D1: number analyzed (Participants) | 24 | 9
  Fear of Future Health: Change at C5 D1 | 0.00 (35.44) | 14.81 (29.40)
  Ability to Plan Future: Change at C5 D1: number analyzed (Participants) | 25 | 9
  Ability to Plan Future: Change at C5 D1 | 20.00 (41.94) | -11.11 (16.67)
  Pancreatic Pain: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Pancreatic Pain: Change at C6 D1 | -3.76 (24.06) | -12.50 (30.81)
  Eating Related Items: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Eating Related Items: Change at C6 D1 | -4.90 (50.95) | 8.33 (21.52)
  Altered Bowel Habits: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Altered Bowel Habits: Change at C6 D1 | 13.73 (25.16) | -8.33 (28.87)
  Jaundice: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Jaundice: Change at C6 D1 | 1.96 (11.61) | -16.67 (45.13)
  Body Image: Change at C6 D1: number analyzed (Participants) | 16 | 4
  Body Image: Change at C6 D1 | 23.96 (31.60) | 0.00 (0.00)
  Health Care Satisfaction: Change at C6 D1: number analyzed (Participants) | 16 | 4
  Health Care Satisfaction: Change at C6 D1 | -11.46 (42.04) | -25.00 (21.52)
  Sexual Functioning: Change at C6 D1: number analyzed (Participants) | 13 | 4
  Sexual Functioning: Change at C6 D1 | -7.69 (30.14) | -20.83 (49.77)
  Ascites: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Ascites: Change at C6 D1 | -1.96 (24.92) | -8.33 (31.91)
  Indigestion: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Indigestion: Change at C6 D1 | 3.92 (35.12) | -16.67 (19.25)
  Flatulence: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Flatulence: Change at C6 D1 | 1.96 (27.56) | -8.33 (16.67)
  Cachexia: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Cachexia: Change at C6 D1 | 4.90 (31.05) | -20.83 (15.96)
  Side Effects: Change at C6 D1: number analyzed (Participants) | 17 | 4
  Side Effects: Change at C6 D1 | 16.34 (30.40) | -22.22 (15.71)
  Fear of Future Health: Change at C6 D1: number analyzed (Participants) | 15 | 4
  Fear of Future Health: Change at C6 D1 | -4.44 (45.19) | 0.00 (0.00)
  Ability to Plan Future: Change at C6 D1: number analyzed (Participants) | 16 | 4
  Ability to Plan Future: Change at C6 D1 | 12.50 (54.26) | 16.67 (63.83)
  Pancreatic Pain: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Pancreatic Pain: Change at C7 D1 | -3.70 (22.09) | -16.67 (11.79)
  Eating Related Items: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Eating Related Items: Change at C7 D1 | -14.81 (31.67) | 8.33 (11.79)
  Altered Bowel Habits: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Altered Bowel Habits: Change at C7 D1 | 5.56 (23.57) | 25.00 (58.93)
  Jaundice: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Jaundice: Change at C7 D1 | 5.56 (11.79) | -41.67 (58.93)
  Body Image: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Body Image: Change at C7 D1 | 16.67 (41.67) | -25.00 (58.93)
  Health Care Satisfaction: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Health Care Satisfaction: Change at C7 D1 | 5.56 (26.35) | -33.33 (0.00)
  Sexual Functioning: Change at C7 D1: number analyzed (Participants) | 7 | 2
  Sexual Functioning: Change at C7 D1 | -9.52 (18.90) | -41.67 (11.79)
  Ascites: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Ascites: Change at C7 D1 | 0.00 (0.00) | 0.00 (0.00)
  Indigestion: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Indigestion: Change at C7 D1 | -7.41 (22.22) | 0.00 (0.00)
  Flatulence: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Flatulence: Change at C7 D1 | -3.70 (30.93) | -16.67 (23.57)
  Cachexia: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Cachexia: Change at C7 D1 | 5.56 (25.00) | -8.33 (35.36)
  Side Effects: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Side Effects: Change at C7 D1 | 8.64 (25.93) | -22.22 (31.43)
  Fear of Future Health: Change at C7 D1: number analyzed (Participants) | 8 | 2
  Fear of Future Health: Change at C7 D1 | 4.17 (27.82) | -16.67 (70.71)
  Ability to Plan Future: Change at C7 D1: number analyzed (Participants) | 9 | 2
  Ability to Plan Future: Change at C7 D1 | 14.81 (55.56) | 33.33 (47.14)
  Pancreatic Pain: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Pancreatic Pain: Change at C8 D1 | -1.54 (25.99) | -25.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Eating Related Items: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Eating Related Items: Change at C8 D1 | 3.70 (48.43) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Altered Bowel Habits: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Altered Bowel Habits: Change at C8 D1 | 14.81 (22.74) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Jaundice: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Jaundice: Change at C8 D1 | 9.26 (12.11) | -83.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Body Image: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Body Image: Change at C8 D1 | 22.22 (37.27) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Health Care Satisfaction: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Health Care Satisfaction: Change at C8 D1 | 3.70 (27.36) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Sexual Functioning: Change at C8 D1: number analyzed (Participants) | 7 | 1
  Sexual Functioning: Change at C8 D1 | -7.14 (13.11) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ascites: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Ascites: Change at C8 D1 | -3.70 (26.06) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Indigestion: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Indigestion: Change at C8 D1 | -7.41 (40.06) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Flatulence: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Flatulence: Change at C8 D1 | -11.11 (33.33) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cachexia: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Cachexia: Change at C8 D1 | 11.11 (26.35) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Side Effects: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Side Effects: Change at C8 D1 | 11.11 (35.14) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fear of Future Health: Change at C8 D1: number analyzed (Participants) | 8 | 1
  Fear of Future Health: Change at C8 D1 | 4.17 (45.21) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ability to Plan Future: Change at C8 D1: number analyzed (Participants) | 9 | 1
  Ability to Plan Future: Change at C8 D1 | 11.11 (64.55) | 66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pancreatic Pain: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Pancreatic Pain: Change at C9 D1 | 0.00 (30.43) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Eating Related Items: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Eating Related Items: Change at C9 D1 | 14.29 (39.00) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Altered Bowel Habits: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Altered Bowel Habits: Change at C9 D1 | 23.81 (25.20) | -50.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Jaundice: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Jaundice: Change at C9 D1 | 9.52 (16.27) | -66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Body Image: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Body Image: Change at C9 D1 | 28.57 (35.63) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Health Care Satisfaction: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Health Care Satisfaction: Change at C9 D1 | 2.38 (24.40) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Sexual Functioning: Change at C9 D1: number analyzed (Participants) | 5 | 1
  Sexual Functioning: Change at C9 D1 | -13.33 (29.81) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ascites: Change at C9 D1: number analyzed (Participants) | 6 | 1
  Ascites: Change at C9 D1 | -11.11 (34.43) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Indigestion: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Indigestion: Change at C9 D1 | 4.76 (35.63) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Flatulence: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Flatulence: Change at C9 D1 | 14.29 (26.23) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cachexia: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Cachexia: Change at C9 D1 | 23.81 (34.50) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Side Effects: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Side Effects: Change at C9 D1 | 31.75 (33.60) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fear of Future Health: Change at C9 D1: number analyzed (Participants) | 6 | 1
  Fear of Future Health: Change at C9 D1 | -16.67 (40.82) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ability to Plan Future: Change at C9 D1: number analyzed (Participants) | 7 | 1
  Ability to Plan Future: Change at C9 D1 | 19.05 (42.41) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pancreatic Pain: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Pancreatic Pain: Change at C10 D1 | 8.33 (25.28) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Eating Related Items: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Eating Related Items: Change at C10 D1 | 25.00 (25.28) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Altered Bowel Habits: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Altered Bowel Habits: Change at C10 D1 | 27.78 (22.77) | -50.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Jaundice: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Jaundice: Change at C10 D1 | 2.78 (16.39) | -83.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Body Image: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Body Image: Change at C10 D1 | 25.00 (29.34) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Health Care Satisfaction: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Health Care Satisfaction: Change at C10 D1 | 13.89 (30.58) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Sexual Functioning: Change at C10 D1: number analyzed (Participants) | 5 | 1
  Sexual Functioning: Change at C10 D1 | -13.33 (29.81) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ascites: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Ascites: Change at C10 D1 | 0.00 (21.08) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Indigestion: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Indigestion: Change at C10 D1 | 27.78 (25.09) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Flatulence: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Flatulence: Change at C10 D1 | 16.67 (18.26) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cachexia: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Cachexia: Change at C10 D1 | 25.00 (39.09) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Side Effects: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Side Effects: Change at C10 D1 | 37.04 (28.69) | 11.11 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fear of Future Health: Change at C10 D1: number analyzed (Participants) | 5 | 1
  Fear of Future Health: Change at C10 D1 | 0.00 (0.00) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ability to Plan Future: Change at C10 D1: number analyzed (Participants) | 6 | 1
  Ability to Plan Future: Change at C10 D1 | 33.33 (42.16) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pancreatic Pain: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Pancreatic Pain: Change at C11 D1 | 5.56 (47.39) | -8.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Eating Related Items: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Eating Related Items: Change at C11 D1 | 38.89 (53.58) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Altered Bowel Habits: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Altered Bowel Habits: Change at C11 D1 | 50.00 (44.10) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Jaundice: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Jaundice: Change at C11 D1 | 16.67 (44.10) | -83.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Body Image: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Body Image: Change at C11 D1 | 50.00 (44.10) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Health Care Satisfaction: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Health Care Satisfaction: Change at C11 D1 | 27.78 (25.46) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Sexual Functioning: Change at C11 D1: number analyzed (Participants) | 2 | 1
  Sexual Functioning: Change at C11 D1 | -33.33 (47.14) | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ascites: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Ascites: Change at C11 D1 | 22.22 (38.49) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Indigestion: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Indigestion: Change at C11 D1 | 11.11 (19.25) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Flatulence: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Flatulence: Change at C11 D1 | 11.11 (19.25) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cachexia: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Cachexia: Change at C11 D1 | 55.56 (25.46) | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Side Effects: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Side Effects: Change at C11 D1 | 55.56 (50.92) | 11.11 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fear of Future Health: Change at C11 D1: number analyzed (Participants) | 2 | 1
  Fear of Future Health: Change at C11 D1 | 0.00 (0.00) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ability to Plan Future: Change at C11 D1: number analyzed (Participants) | 3 | 1
  Ability to Plan Future: Change at C11 D1 | 44.44 (50.92) | 66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Pancreatic Pain: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Pancreatic Pain: Change at C12 D1 | -5.56 (20.97) |
  Eating Related Items: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Eating Related Items: Change at C12 D1 | 16.67 (16.67) |
  Altered Bowel Habits: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Altered Bowel Habits: Change at C12 D1 | 27.78 (34.69) |
  Jaundice: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Jaundice: Change at C12 D1 | 0.00 (0.00) |
  Body Image: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Body Image: Change at C12 D1 | 16.67 (16.67) |
  Health Care Satisfaction: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Health Care Satisfaction: Change at C12 D1 | -5.56 (41.94) |
  Sexual Functioning: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Sexual Functioning: Change at C12 D1 | 0.00 (66.67) |
  Ascites: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Ascites: Change at C12 D1 | -22.22 (19.25) |
  Indigestion: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Indigestion: Change at C12 D1 | 0.00 (0.00) |
  Flatulence: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Flatulence: Change at C12 D1 | 0.00 (0.00) |
  Cachexia: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Cachexia: Change at C12 D1 | 33.33 (28.87) |
  Side Effects: Change at C12 D1(n=3,0): number analyzed (Participants) | 3 | 0
  Side Effects: Change at C12 D1(n=3,0) | 33.33 (40.06) |
  Fear of Future Health: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Fear of Future Health: Change at C12 D1 | 0.00 (0.00) |
  Ability to Plan Future: Change at C12 D1: number analyzed (Participants) | 3 | 0
  Ability to Plan Future: Change at C12 D1 | 0.00 (0.00) |
  Pancreatic Pain: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Pancreatic Pain: Change at C13 D1 | 20.83 (5.89) |
  Eating Related Items: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Eating Related Items: Change at C13 D1 | 58.33 (58.93) |
  Altered Bowel Habits: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Altered Bowel Habits: Change at C13 D1 | 8.33 (11.79) |
  Jaundice: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Jaundice: Change at C13 D1 | 25.00 (35.36) |
  Body Image: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Body Image: Change at C13 D1 | 41.67 (58.93) |
  Health Care Satisfaction: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Health Care Satisfaction: Change at C13 D1 | -16.67 (23.57) |
  Sexual Functioning: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Sexual Functioning: Change at C13 D1 | -50.00 (23.57) |
  Ascites: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Ascites: Change at C13 D1 | 16.67 (23.57) |
  Indigestion: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Indigestion: Change at C13 D1 | 0.00 (0.00) |
  Flatulence: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Flatulence: Change at C13 D1 | 16.67 (23.57) |
  Cachexia: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Cachexia: Change at C13 D1 | 33.33 (47.14) |
  Side Effects: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Side Effects: Change at C13 D1 | 16.67 (7.86) |
  Fear of Future Health: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Fear of Future Health: Change at C13 D1 | 0.00 (0.00) |
  Ability to Plan Future: Change at C13 D1: number analyzed (Participants) | 2 | 0
  Ability to Plan Future: Change at C13 D1 | 16.67 (23.57) |
  Pancreatic Pain: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Pancreatic Pain: Change at C14 D1 | -8.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Eating Related Items: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Eating Related Items: Change at C14 D1 | 16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Altered Bowel Habits: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Altered Bowel Habits: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Jaundice: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Jaundice: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Body Image: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Body Image: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Health Care Satisfaction: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Health Care Satisfaction: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Sexual Functioning: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Sexual Functioning: Change at C14 D1 | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Ascites: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Ascites: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Indigestion: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Indigestion: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Flatulence: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Flatulence: Change at C14 D1 | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Cachexia: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Cachexia: Change at C14 D1 | 50.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Side Effects: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Side Effects: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Fear of Future Health: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Fear of Future Health: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Ability to Plan Future: Change at C14 D1: number analyzed (Participants) | 1 | 0
  Ability to Plan Future: Change at C14 D1 | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. |
  Pancreatic Pain: Change at EoS: number analyzed (Participants) | 2 | 1
  Pancreatic Pain: Change at EoS | 58.33 (35.36) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Eating Related Items: Change at EoS: number analyzed (Participants) | 2 | 1
  Eating Related Items: Change at EoS | 25.00 (82.50) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Altered Bowel Habits: Change at EoS: number analyzed (Participants) | 2 | 1
  Altered Bowel Habits: Change at EoS | 83.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Jaundice: Change at EoS: number analyzed (Participants) | 2 | 1
  Jaundice: Change at EoS | 8.33 (11.79) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Body Image: Change at EoS: number analyzed (Participants) | 2 | 1
  Body Image: Change at EoS | 66.67 (0.00) | -16.67 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Health Care Satisfaction: Change at EoS: number analyzed (Participants) | 1 | 1
  Health Care Satisfaction: Change at EoS | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Sexual Functioning: Change at EoS: number analyzed (Participants) | 1 | 1
  Sexual Functioning: Change at EoS | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable. | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ascites: Change at EoS: number analyzed (Participants) | 2 | 1
  Ascites: Change at EoS | 33.33 (47.14) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Indigestion: Change at EoS: number analyzed (Participants) | 2 | 1
  Indigestion: Change at EoS | 33.33 (47.14) | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Flatulence: Change at EoS: number analyzed (Participants) | 2 | 1
  Flatulence: Change at EoS | 83.33 (23.57) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Cachexia: Change at EoS: number analyzed (Participants) | 2 | 1
  Cachexia: Change at EoS | 66.67 (0.00) | 0.00 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Side Effects: Change at EoS: number analyzed (Participants) | 2 | 1
  Side Effects: Change at EoS | 19.44 (90.35) | -11.11 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Fear of Future Health: Change at EoS: number analyzed (Participants) | 1 | 1
  Fear of Future Health: Change at EoS | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable. | -33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
  Ability to Plan Future: Change at EoS: number analyzed (Participants) | 1 | 1
  Ability to Plan Future: Change at EoS | 66.67 (NA) — Standard deviation was not calculated because only one participant was evaluable. | 33.33 (NA) — Standard deviation was not calculated because only one participant was evaluable.
Statistical Analysis 1: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 2.59, 95% CI 2-sided [-10.11 to 15.29]
Statistical Analysis 2: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.41, 95% CI 2-sided [-13.39 to 20.20]
Statistical Analysis 3: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 19.70, 95% CI 2-sided [5.96 to 33.43]
Statistical Analysis 4: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.70, 95% CI 2-sided [0.93 to 24.47]
Statistical Analysis 5: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.10, 95% CI 2-sided [1.28 to 28.91]
Statistical Analysis 6: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 4.36, 95% CI 2-sided [-14.59 to 23.30]
Statistical Analysis 7: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -21.19, 95% CI 2-sided [-37.53 to -4.85]
Statistical Analysis 8: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.82, 95% CI 2-sided [-25.04 to 9.40]
Statistical Analysis 9: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.95, 95% CI 2-sided [-9.59 to 21.50]
Statistical Analysis 10: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.39, 95% CI 2-sided [-1.61 to 30.40]
Statistical Analysis 11: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.50, 95% CI 2-sided [2.78 to 22.22]
Statistical Analysis 12: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.88, 95% CI 2-sided [1.36 to 20.39]
Statistical Analysis 13: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -2.33, 95% CI 2-sided [-16.36 to 11.71]
Statistical Analysis 14: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 2 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 6.21, 95% CI 2-sided [-11.78 to 24.20]
Statistical Analysis 15: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.87, 95% CI 2-sided [0.79 to 28.94]
Statistical Analysis 16: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.49, 95% CI 2-sided [-7.45 to 34.42]
Statistical Analysis 17: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 18.86, 95% CI 2-sided [0.17 to 37.55]
Statistical Analysis 18: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.57, 95% CI 2-sided [0.66 to 22.48]
Statistical Analysis 19: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 18.72, 95% CI 2-sided [0.49 to 36.95]
Statistical Analysis 20: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -10.61, 95% CI 2-sided [-32.40 to 11.17]
Statistical Analysis 21: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [-14.63 to 17.27]
Statistical Analysis 22: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-14.70 to 17.78]
Statistical Analysis 23: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.05, 95% CI 2-sided [-10.65 to 32.75]
Statistical Analysis 24: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.40, 95% CI 2-sided [-17.33 to 24.13]
Statistical Analysis 25: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.27, 95% CI 2-sided [-4.40 to 22.93]
Statistical Analysis 26: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 19.19, 95% CI 2-sided [2.99 to 35.39]
Statistical Analysis 27: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-23.70 to 22.43]
Statistical Analysis 28: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 3 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 21.51, 95% CI 2-sided [-3.10 to 46.12]
Statistical Analysis 29: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.19, 95% CI 2-sided [-21.57 to 13.19]
Statistical Analysis 30: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -12.60, 95% CI 2-sided [-32.86 to 7.66]
Statistical Analysis 31: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.25, 95% CI 2-sided [-10.33 to 34.82]
Statistical Analysis 32: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.84, 95% CI 2-sided [-0.18 to 25.85]
Statistical Analysis 33: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.85, 95% CI 2-sided [-16.45 to 24.14]
Statistical Analysis 34: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 7.05, 95% CI 2-sided [-23.23 to 37.34]
Statistical Analysis 35: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -2.53, 95% CI 2-sided [-26.55 to 21.50]
Statistical Analysis 36: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -9.46, 95% CI 2-sided [-27.48 to 8.56]
Statistical Analysis 37: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -6.96, 95% CI 2-sided [-30.62 to 16.70]
Statistical Analysis 38: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 3.71, 95% CI 2-sided [-20.37 to 27.80]
Statistical Analysis 39: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.04, 95% CI 2-sided [-5.73 to 31.81]
Statistical Analysis 40: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.12, 95% CI 2-sided [-3.23 to 33.46]
Statistical Analysis 41: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.91, 95% CI 2-sided [-36.18 to 20.37]
Statistical Analysis 42: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 4 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.38, 95% CI 2-sided [-20.24 to 51.01]
Statistical Analysis 43: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.25, 95% CI 2-sided [-10.09 to 32.59]
Statistical Analysis 44: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 7.41, 95% CI 2-sided [-25.22 to 40.03]
Statistical Analysis 45: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 28.28, 95% CI 2-sided [4.23 to 52.32]
Statistical Analysis 46: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 24.22, 95% CI 2-sided [5.09 to 43.34]
Statistical Analysis 47: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.11, 95% CI 2-sided [-0.16 to 50.38]
Statistical Analysis 48: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -10.07, 95% CI 2-sided [-47.95 to 27.80]
Statistical Analysis 49: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.61, 95% CI 2-sided [-21.78 to 14.57]
Statistical Analysis 50: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.98, 95% CI 2-sided [-17.02 to 28.99]
Statistical Analysis 51: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.08, 95% CI 2-sided [-5.39 to 49.55]
Statistical Analysis 52: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 9.78, 95% CI 2-sided [-15.33 to 34.89]
Statistical Analysis 53: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 15.81, 95% CI 2-sided [-10.43 to 42.06]
Statistical Analysis 54: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 21.77, 95% CI 2-sided [1.11 to 42.43]
Statistical Analysis 55: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -14.81, 95% CI 2-sided [-41.91 to 12.28]
Statistical Analysis 56: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 5 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 31.11, 95% CI 2-sided [1.60 to 60.62]
Statistical Analysis 57: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 8.74, 95% CI 2-sided [-20.62 to 38.10]
Statistical Analysis 58: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -13.24, 95% CI 2-sided [-68.52 to 42.05]
Statistical Analysis 59: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.06, 95% CI 2-sided [-7.93 to 52.05]
Statistical Analysis 60: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 18.63, 95% CI 2-sided [-5.64 to 42.89]
Statistical Analysis 61: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.96, 95% CI 2-sided [-9.93 to 57.84]
Statistical Analysis 62: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.54, 95% CI 2-sided [-32.70 to 59.78]
Statistical Analysis 63: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.14, 95% CI 2-sided [-29.46 to 55.74]
Statistical Analysis 64: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 6.37, 95% CI 2-sided [-24.04 to 36.79]
Statistical Analysis 65: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.59, 95% CI 2-sided [-17.94 to 59.12]
Statistical Analysis 66: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 10.29, 95% CI 2-sided [-20.12 to 40.71]
Statistical Analysis 67: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.74, 95% CI 2-sided [-8.22 to 59.69]
Statistical Analysis 68: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 38.56, 95% CI 2-sided [5.32 to 71.81]
Statistical Analysis 69: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.44, 95% CI 2-sided [-53.14 to 44.25]
Statistical Analysis 70: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 6 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -4.17, 95% CI 2-sided [-69.90 to 61.57]
Statistical Analysis 71: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.96, 95% CI 2-sided [-24.52 to 50.45]
Statistical Analysis 72: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -23.15, 95% CI 2-sided [-76.41 to 30.11]
Statistical Analysis 73: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -19.44, 95% CI 2-sided [-71.89 to 33.00]
Statistical Analysis 74: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 47.22, 95% CI 2-sided [7.31 to 87.13]
Statistical Analysis 75: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 41.67, 95% CI 2-sided [-36.00 to 119.34]
Statistical Analysis 76: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 38.89, 95% CI 2-sided [-5.05 to 82.83]
Statistical Analysis 77: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 32.14, 95% CI 2-sided [-2.09 to 66.37]
Statistical Analysis 78: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.41, 95% CI 2-sided [-44.46 to 29.64]
Statistical Analysis 79: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 12.96, 95% CI 2-sided [-40.45 to 66.37]
Statistical Analysis 80: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.89, 95% CI 2-sided [-32.71 to 60.49]
Statistical Analysis 81: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 30.86, 95% CI 2-sided [-16.16 to 77.89]
Statistical Analysis 82: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.83, 95% CI 2-sided [-44.95 to 86.62]
Statistical Analysis 83: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 7 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -18.52, 95% CI 2-sided [-115.22 to 78.19]
Statistical Analysis 84: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.46, 95% CI 2-sided [-39.71 to 86.63]
Statistical Analysis 85: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -12.96, 95% CI 2-sided [-130.69 to 104.76]
Statistical Analysis 86: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 48.15, 95% CI 2-sided [-7.12 to 103.42]
Statistical Analysis 87: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 92.59, 95% CI 2-sided [63.16 to 122.02]
Statistical Analysis 88: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [-85.03 to 96.14]
Statistical Analysis 89: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 37.04, 95% CI 2-sided [-29.46 to 103.54]
Statistical Analysis 90: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.14, 95% CI 2-sided [-41.45 to 27.16]
Statistical Analysis 91: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-67.04 to 59.64]
Statistical Analysis 92: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -7.41, 95% CI 2-sided [-104.79 to 89.97]
Statistical Analysis 93: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 22.22, 95% CI 2-sided [-58.80 to 103.25]
Statistical Analysis 94: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.78, 95% CI 2-sided [-36.28 to 91.83]
Statistical Analysis 95: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.11, 95% CI 2-sided [-74.30 to 96.52]
Statistical Analysis 96: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -29.17, 95% CI 2-sided [-142.55 to 84.21]
Statistical Analysis 97: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 8 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -55.56, 95% CI 2-sided [-212.46 to 101.35]
Statistical Analysis 98: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.67, 95% CI 2-sided [-62.93 to 96.26]
Statistical Analysis 99: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.29, 95% CI 2-sided [-87.74 to 116.31]
Statistical Analysis 100: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 73.81, 95% CI 2-sided [7.90 to 139.72]
Statistical Analysis 101: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 76.19, 95% CI 2-sided [33.64 to 118.74]
Statistical Analysis 102: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 28.57, 95% CI 2-sided [-64.64 to 121.79]
Statistical Analysis 103: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 35.71, 95% CI 2-sided [-28.11 to 99.53]
Statistical Analysis 104: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -13.33, 95% CI 2-sided [-104.01 to 77.34]
Statistical Analysis 105: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -44.44, 95% CI 2-sided [-140.03 to 51.14]
Statistical Analysis 106: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 4.76, 95% CI 2-sided [-88.45 to 97.98]
Statistical Analysis 107: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 14.29, 95% CI 2-sided [-54.32 to 82.89]
Statistical Analysis 108: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 23.81, 95% CI 2-sided [-66.45 to 114.07]
Statistical Analysis 109: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 31.75, 95% CI 2-sided [-56.14 to 119.63]
Statistical Analysis 110: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in fear of future health at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -50.00, 95% CI 2-sided [-163.35 to 63.35]
Statistical Analysis 111: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 9 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -14.29, 95% CI 2-sided [-125.23 to 96.66]
Statistical Analysis 112: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [-45.18 to 95.18]
Statistical Analysis 113: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [-45.18 to 95.18]
Statistical Analysis 114: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 77.78, 95% CI 2-sided [14.55 to 141.00]
Statistical Analysis 115: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 86.11, 95% CI 2-sided [40.61 to 131.61]
Statistical Analysis 116: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [-56.48 to 106.48]
Statistical Analysis 117: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 47.22, 95% CI 2-sided [-37.69 to 132.13]
Statistical Analysis 118: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 20.00, 95% CI 2-sided [-70.68 to 110.68]
Statistical Analysis 119: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -33.33, 95% CI 2-sided [-91.87 to 25.20]
Statistical Analysis 120: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 27.78, 95% CI 2-sided [-41.89 to 97.45]
Statistical Analysis 121: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 16.67, 95% CI 2-sided [-34.03 to 67.36]
Statistical Analysis 122: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 8.33, 95% CI 2-sided [-100.19 to 116.86]
Statistical Analysis 123: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.93, 95% CI 2-sided [-53.73 to 105.58]
Statistical Analysis 124: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 10 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-117.07 to 117.07]
Statistical Analysis 125: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 13.89, 95% CI 2-sided [-221.53 to 249.31]
Statistical Analysis 126: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 5.56, 95% CI 2-sided [-260.62 to 271.74]
Statistical Analysis 127: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 66.67, 95% CI 2-sided [-152.41 to 285.75]
Statistical Analysis 128: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 100.00, 95% CI 2-sided [-119.08 to 319.08]
Statistical Analysis 129: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in body image at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 33.33, 95% CI 2-sided [-185.75 to 252.41]
Statistical Analysis 130: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in health care satisfaction at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 44.44, 95% CI 2-sided [-82.04 to 170.93]
Statistical Analysis 131: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in sexual functioning at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-733.59 to 733.59]
Statistical Analysis 132: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -11.11, 95% CI 2-sided [-202.34 to 180.12]
Statistical Analysis 133: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.11, 95% CI 2-sided [-84.50 to 106.73]
Statistical Analysis 134: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 11.11, 95% CI 2-sided [-84.50 to 106.73]
Statistical Analysis 135: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in cachexia at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 38.89, 95% CI 2-sided [-87.60 to 165.37]
Statistical Analysis 136: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 44.44, 95% CI 2-sided [-208.53 to 297.42]
Statistical Analysis 137: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ability to plan future at Cycle 11 Day 1, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = -22.22, 95% CI 2-sided [-275.19 to 230.75]
Statistical Analysis 138: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in pancreatic pain at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 58.33, 95% CI 2-sided [-491.86 to 608.53]
Statistical Analysis 139: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in eating related items at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 25.00, 95% CI 2-sided [-1258.79 to 1308.79]
Statistical Analysis 140: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in altered bowel habits at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 83.33, 95% CI 2-sided [-283.46 to 450.13]
Statistical Analysis 141: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in jaundice at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 8.33, 95% CI 2-sided [-175.06 to 191.73]
Statistical Analysis 142: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in ascites at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-733.59 to 733.59]
Statistical Analysis 143: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in indigestion at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-733.59 to 733.59]
Statistical Analysis 144: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in flatulence at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 83.33, 95% CI 2-sided [-283.46 to 450.13]
Statistical Analysis 145: Comparison: Axitinib + Gemcitabine vs Gemcitabine; For change in side effects at EoS, mean change difference was used to compare the two treatment groups; Test type: Superiority or Other; Mean Difference (Final Values) = 30.56, 95% CI 2-sided [-1375.5 to 1436.61]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Axitinib + Gemcitabine: Axitinib (AG-013736) 5 mg tablet orally twice daily (BID) from Day 1 of Cycle 1 (28 days) and all subsequent cycles (28 days). Gemcitabine 1000 mg/m^2 30-minute infusion on Day 1, 8 and 15 of each cycle.
Arm/Group | Axitinib + Gemcitabine (Phase 1 Lead-In) | Axitinib + Gemcitabine | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 3/8 | 35/68 | 10/31
Other Adverse Events (participants affected / at risk) | 7/8 | 67/68 | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Gemcitabine (Phase 1 Lead-In) (N=8) | Axitinib + Gemcitabine (N=68) | Gemcitabine (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 4 | 0
Chest pain (General disorders) | 0 | 1 | 0
Device occlusion (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 6 | 0
Fatigue (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Lung abscess (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Gemcitabine (Phase 1 Lead-In) (N=8) | Axitinib + Gemcitabine (N=68) | Gemcitabine (N=31)
Anaemia (Blood and lymphatic system disorders) | 4 | 16 | 7
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 15 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 10 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 16 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 11 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 3 | 5
Constipation (Gastrointestinal disorders) | 2 | 18 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 35 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 5 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 9 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 5 | 2
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 5 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 30 | 15
Oral pain (Gastrointestinal disorders) | 0 | 6 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 12 | 2
Tongue coated (Gastrointestinal disorders) | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 29 | 12
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 22 | 4
Catheter site pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 5 | 0
Chills (General disorders) | 0 | 5 | 3
Device occlusion (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 7 | 29 | 10
Feeling cold (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 1 | 0
Mucosal dryness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 3 | 12 | 2
Oedema (General disorders) | 0 | 6 | 0
Oedema peripheral (General disorders) | 1 | 11 | 8
Pain (General disorders) | 0 | 10 | 2
Performance status decreased (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 12 | 7
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 3 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gingival abscess (Infections and infestations) | 1 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0
Periodontal infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 9 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Aspartate aminotransferase (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood albumin increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase (Investigations) | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 3 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Haemoglobin (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 5 | 2
Heart rate increased (Investigations) | 0 | 0 | 1
International normalised ratio (Investigations) | 0 | 0 | 1
Neutrophil count (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 4 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 2 | 1
Weight decreased (Investigations) | 1 | 16 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 29 | 10
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 11 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 12 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 8 | 3
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 7 | 2
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 9 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 5 | 0
Lethargy (Nervous system disorders) | 0 | 6 | 0
Neuropathy (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 1
Sensory loss (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 9 | 3
Confusional state (Psychiatric disorders) | 0 | 2 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 7 | 2
Insomnia (Psychiatric disorders) | 2 | 6 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 6 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 15 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 10 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 12 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pancreaticoduodenectomy (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 4 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 16 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Population pharmacokinetics was not presented, as the data was not available for the single study and data of other axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.